CLINICAL TRIAL: NCT00428779
Title: Neuromuscular and Cognitive Fatigue During a 24h Treadmill Running Exercise.
Brief Title: Neuromuscular and Cognitive Fatigue During a 24 Hour Treadmill Running Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, CHU de Saint-Etienne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0601095; DGS 2006-0111; 2006-A00312-49
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Running during 24 hours; Voluntary evoked force on the muscles; Electrically evoked force on the muscles; EMG activity; Muscle biopsy; subjects will be recruited among experienced ultra-runners
MeSH Terms: interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients running during 24 hours without sleep
  Interventions: Procedure: running during 24 hours without sleep
- 2 (Placebo Comparator): patients without sleep during 24 hours
  Interventions: Other: no sleeping

INTERVENTIONS:
Procedure: running during 24 hours without sleep — patients running during 24 hours without sleep
  Arms: 1
Other: no sleeping — patients without sleep during 24 hours
  Arms: 2

SUMMARY:
The main purpose of the present study is to determine the relative contributions of central and peripheral fatigue during an ultra-endurance exercise.

DETAILED DESCRIPTION:
For that purpose, 14 subjects running 24 hours on a treadmill will be compared with a control group being awake during the same period. Subjects who running will have electrically evoked forces on the muscles associated EMG activity, blood samples and muscle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* The subjects of the experimental group will be recruited among experienced ultra-runners . They all have run at least a 12 hour race or longer.
* The control group will be recruited among experienced ultra-runners . Age of control group will be age experimental group more or less 2 years.

Exclusion Criteria:

* The subjects will not be selected if:

  * they were injured in the 3 months before the experiment
  * they had a tendon or joint pathology that could impair strength measurements.
  * they participate to an other experiment at the same time

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
-Voluntary and electrically evoked forces on the contracted muscles | 24 hours

SECONDARY OUTCOMES:
Electrically evoked forces on the relaxed muscles and associated EMG activity | 24 hours
Blood samples before the exercise | every 4 hours
Muscle biopsy (vastus lateralis) | before and after the exercise

CONTACTS AND LOCATIONS:
Overall Officials: DENIS Christian, Professor, Study Chair — Service de médecine du sport, CHU SAINT-ETIENNE
Locations (1):
- Pr André GEYSSANT, Saint-Etienne, France

REFERENCES:
- [Result] Morin JB, Samozino P, Feasson L, Geyssant A, Millet G. Effects of muscular biopsy on the mechanics of running. Eur J Appl Physiol. 2009 Jan;105(2):185-90. doi: 10.1007/s00421-008-0888-2. Epub 2008 Oct 8. PMID 18841378
- [Derived] Jamart C, Francaux M, Millet GY, Deldicque L, Frere D, Feasson L. Modulation of autophagy and ubiquitin-proteasome pathways during ultra-endurance running. J Appl Physiol (1985). 2012 May;112(9):1529-37. doi: 10.1152/japplphysiol.00952.2011. Epub 2012 Feb 16. PMID 22345427